



# "CASCADES" CLINICAL TRIAL PROTOCOL SUMMARY

"A randomized, open-label, clinical trial evaluating the anti-atherosclerotic efficacy of selected antidiabetic drugs in patients with coronary artery disease and pre-diabetic conditions. CASCADES

Trial"



**Date and version number** Version 2.1 dated 06/09/2024

Protocol symbol CSDS.IV/VIII/2023

**EU CT number** 2023-508525-27-00

Type of test non-commercial clinical trial

Center Cardinal Stefan Wyszyński National Institute of Cardiology –

National Research Institute

**Principal investigator** dr n. med Jan Henzel

Clinic of Coronary Artery Disease and Structural Heart Diseases – National Research Institute, ul. Alpejska 42, 04-628 Warsaw, tel.

+48 22 343-43-42

Sponsor Cardinal Stefan Wyszyński National Institute of Cardiology –

National Research Institute, ul. Alpejska 42, 04-628 Warsaw, tel.

+48 22 343-43-42

**Funding organization** Medical Research Agency, ul. Stanisława Moniuszki 1A, 00-014

Warsaw

**Project management** Clinical Research Support Center, Cardinal Stefan Wyszyński

National Institute of Cardiology – National Research Institute, 42

Alpejska St., 04-628 Warsaw, tel. +48 22 343-40-80; e-mail:

kkotlinska@ikard.pl



| Study title | A randomized, open-label, clinical trial evaluating the anti-<br>atherosclerotic efficacy of selected antidiabetic drugs |
|---|---|
| | atherosclerotic efficacy of selected antidiabetic drugs in patients with coronary artery disease and pre-diabetic |
| | conditions. CASCADES Trial. |
| Acronym | CASCADES |
| EU CT: | 2023-508525-27 |
| Sponsor | Cardinal Stefan Wyszyński National Institute of Cardiology – National Research Institute, ul. Alpejska 42, 04-628 Warsaw. |
| Researcher | dr n. med. Jan Henzel, Department of Coronary Artery Disease and Structural Heart Diseases, Cardinal Stefan Wyszyński National Institute of Cardiology – National Research Institute, ul. Alpejska 42, 04-628 |
| | Warsaw, tel. 22 343 34 42, e-mail: jhenzel@ikard.pl |
| Research center | Cardinal Stefan Wyszyński National Institute of Cardiology – National Research Institute, ul. Alpejska 42, 04-628 Warsaw. Single-center study. |
| Study rationale | The purpose of the study is to compare the anti-atherosclerotic efficacy of oral treatment with a GLP-1 analogue (semaglutide) or an SGLT-2 (so-called "flozin") inhibitor (dapagliflozin) versus routine treatment (metformin) in patients with pre-diabetes and diagnosed coronary artery disease at 24 months. The diagnosis of coronary artery disease will be defined as the presence of coronary atherosclerosis confirmed by coronary artery computed tomography (coronary CT). |
| Clinical phase | IV |
| Study<br>methodology | Randomized controlled, open, with two arms of therapeutic intervention |
| Measurements and procedures | Evaluation of coronary arteries by computed tomography scanning of coronary arteries with contrast Pharmacological intervention: flozin 10 mg vs. semaglutide 3 mg – 7 mg, 14 mg vs. metformin 500 mg – 1000 mg (1:1:1) Physical examination Laboratory tests (venous blood draw, general urinalysis) Measurement of weight, height, blood pressure Assessment of body composition by bioimpedance Resting 12-lead electrocardiogram Non-pharmacological control of coronary heart disease risk factors (dietary, anti-smoking and appropriate physical activity counseling) |





# Inclusion and exclusion criteria

#### Inclusion criteria:

- Age 18 80
- Diagnosed coronary artery disease (coronary artery stenosis of at least 20% with a reference diameter of >2.5 mm or status after percutaneous coronary revascularization procedure found on coronary CT scan)
- Coronary CT scan performed <3 months after inclusion in the study, at least of good quality
- Pre-diabetic status defined as fasting blood glucose 100-125 mg% or Hba1c 5.70-6.49% (measurement documented at the screening/randomization appointment or within 30 days prior to the screening/randomization appointment) or documented, positive result of an oral glucose load test (fasting blood glucose 100-125 mg% and 140-199 mg% 2h after a 75 g oral glucose load) performed up to 30 days before the screening/randomization appointment
- Stable treatment and control of cardiovascular risk factors, including dietary and lifestyle management for at least 4 weeks
- Willing and able to give informed consent to participate in the study
- Willing and able, according to the researcher, to comply with all the requirements of the study

# **Exclusion criteria:**

- Severe valvular defect
- Clinical condition requiring surgical treatment of coronary artery disease
- Status after coronary artery bypass surgery
- Diagnosed diabetes or Hba1c>=6.5% at screening/randomization appointment
- Other severe medical conditions requiring scheduled hospital treatment at the time of the study
- Severe musculoskeletal conditions requiring specific rehabilitation recommendations
- Diagnosed heart failure
- Presence of an artificial valve, cardiac pacing system or other implantable device (such as a cardioverter defibrillator)





| • | Severe arrhy | /thmia/unex | plained loss | of consciousness |
|---|--------------|-------------|--------------|------------------|
|---|--------------|-------------|--------------|------------------|

- Other contraindications to physical activity
- No consent to participate in the study
- Use of glucose-lowering drugs other than metformin
- Use of weight-loss drugs
- Condition after bariatric surgery
- Diagnosed liver disease or ALT, AST above three times the upper limit of normal at screening appointment
- Uncompensated hyperthyroidism
- Pancreatic cancer
- Medullary thyroid cancer
- History of anaphylactic shock after iodine contrast administration
- Chronic kidney disease (eGFR <45 ml/min/1.73 m2)</li>
- History of pancreatitis or active pancreatitis
- Body mass index (BMI) >40 kg/m2
- Pregnancy/lactation
- Participation in another clinical trial
- Other known contraindications to treatment with metformin, dapagliflozin or semaglutide

#### Sample size

### 300 patients

# **Statistical issues**

The study is exploratory, and the primary analysis is designed to separately compare each of the two active groups (treatment: semaglutide or dapagliflozin) with the control group (routine treatment – metformin). According to the scientific literature, the size of the study group was calculated based on a separate comparison of each active group with the control group, without adjusting the power ratios (https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7534018/).

We hypothesized that the % change in the volume of non-calcified atherosclerotic plaque (final values versus initial values) in each active group differed from the control group.

To determine the sample size, the following assumptions were made about treatment efficacy as measured by % change in non-calcified plaque volume compared to baseline values:

Standard deviation of 2.5% for the primary variable.

Treatment difference of at least 1.2% in non-calcified plaque in favor of each study drug compared with the control group.





| Planned study<br>duration | follow-up CT scan at month 2 (282 after withdrawals), with dapagliflozin group, and 93 i 0.90 with a two-sided alpha less Single participant observation Project start date 01/09/2023 Enrolment start date 01/06/2 Completion of treatment and Project completion date 01/0 | n period: 24 months 8 2024 observation 01/06/2028 | participants<br>o, 93 in the |
|---|---|---|---|
| Planned | 01/06/2024 – 01/06/2026 | | |
| enrolment | | | |
| period | _ | Γ | T |
| | Purposes | Endpoints | Time<br>points |
| Co-primary | Evaluation of the effect of GLP-1 analogue treatment on coronary artery disease progression Evaluation of the effect of flozin treatment on the progression of coronary artery disease | Change in % volume of non-calcified atherosclerotic plaque in the coronary arteries assessed by coronary CT versus routine management (intention-to-treat) Change in % volume of non-calcified atherosclerotic plaque in the coronary arteries assessed by coronary CT versus routine management (intention-to-treat) | 24 months 24 months |



| C | F -1 -1: | | <u> </u> |
|---|---|---|---|
| Secondary | Evaluation of the effect of each of the tested drugs vs. control group on progression of coronary artery disease | % change in volume of non-<br>calcified atherosclerotic<br>plaque assessed by<br>coronary CT (as treated)<br>between baseline and end<br>of study | 24 months |
| | Comparison of the effect of semaglutide vs. flozin on coronary artery disease progression | % change in volume of non-<br>calcified atherosclerotic<br>plaque assessed<br>by coronary CT (intention to<br>treat/as treated) between<br>baseline and end of study | 24 months |
| | Evaluation of the effect of each study drug vs. control group/comparison of the effect of semaglutide vs. flozin on progression of coronary artery disease | % change in volume of the entire atherosclerotic plaque assessed by coronary CT) (intention to treat/as treated) between baseline and end of study | 24 months |
| | Evaluation of the effect of each of the tested drugs vs. control group/comparison of the effect of semaglutide vs. flozin on progression of coronary artery disease | % change in volume of individual components of atherosclerotic plaque assessed by coronary CT (intention to treat/as treated) between baseline and end of study | 24 months |
| | Evaluation of the effect of each of the tested drugs vs. control group/comparison of the effect of semaglutide vs. flozin on progression of coronary artery disease | Conversion of non-calcified plaque to calcified plaque (change in % volume of calcified plaque relative to % volume of non-calcified plaque) assessed by coronary CT (intention to treat/as treated) between baseline and end of study | 24 months |



| Evaluation of the effect of each of the tested drugs vs. control group/comparison of the effect of semaglutide vs. flozin on CV risk expressed as the dynamics of high-risk features | 1. Change in the number of high-risk atherosclerotic lesions defined as the presence of at least 2 high-risk features among: - Spotty calcifications - Low attenuation plaques (low attenuation plaque), i.e. plaque density < 30 HU - positive remodeling - napkin ring sign assessed by coronary TK (intention-to-treat/as treated) between baseline and end of study; | 24 months |
|---|---|---|
| | 2. Change in the Pericoronary Fat Attenuation Index assessed by coronary TK (intentionto-treat/as treated) between baseline and end of study | |
| Evaluation of weight change, including body composition, in patients treated with semaglutide vs. patients treated with flozin | <ul> <li>weight</li> <li>body mass index (BMI).</li> <li>fat mass</li> <li>skeletal muscle mass</li> <li>Fat-To-Muscle Ratio (FMR).</li> <li>Body Cell Mass (BCM)</li> <li>Visceral Fat Area (VFA)</li> </ul> | 24 months |
| Evaluation of waist-to-hip index (WHI) change in patients treated with semaglutide vs. patients treated with phlorizin | Change in waist-to-hip index<br>(WHI) between baseline and<br>end of study | 24 months |
| Evaluation of change in inflammatory parameters in patients treated with semaglutide vs. patients treated with phlorizin | Concentration of hsCRP | 24 months |



| Evaluation of change in lipid levels in patients treated with semaglutide vs. patients treated with flozin | <ul> <li>total cholesterol concentration</li> <li>low-density lipoproteins</li> <li>(LDL) concentration</li> <li>high-density lipoproteins</li> <li>(HDL) concentration</li> <li>non-HDL cholesterol concentration</li> <li>triglycerides concentration</li> <li>lipoprotein A concentration</li> </ul> | 24 months |
|---|---|---|
| Evaluation of change in the percentage of glycated hemoglobin (HBA1c) in patients treated with semaglutide vs. patients treated with flozin | Change in the percentage of glycated hemoglobin (HBA1c) between baseline and end of study | 24 months |
| Evaluation of change in the percentage of patients with normal blood pressure in patients treated with semaglutide vs. patients treated with flozin | Change in percentage of patients with normal blood pressure defined as systolic pressure <140 mmHg and diastolic pressure <90 mmHg between baseline and end of study | 24 months |
| Evaluation of change in the percentage of patients currently smoking tobacco or electronic cigarettes in patients treated with semaglutide vs. patients treated with flozin | Change in the percentage of patients currently smoking tobacco (cigarettes, pipe, cigar, tobacco heating products) or electronic cigarettes as defined in section 8.7.a between baseline and end of study | 24 months |
| Evaluation of compliance with physical activity recommendations in patients treated with semaglutide vs. patients treated with flozin | <ul> <li>Percentage of patients classified in the "high" physical activity category;</li> <li>Percentage of patients classified in the "sufficient" physical activity category;</li> </ul> | 24 months |



| Evaluation of dietary compliance in patients treated with semaglutide vs. patients treated with flozin | - Percentage of patients classified in the "insufficient" physical activity category Change in the DASH Index between baseline and end of study | 24 months |
|---|---|---|
| Type 2 diabetes diagnosis | Number of patients diagnosed with diabetes-based on the criteria of the Polish Diabetes Association | 24 months |
| Evaluation of the onset of heart failure requiring hospitalization | Number of hospitalized patients for heart failure | 24 months |
| Number of unplanned hospitalizations | Number of unplanned hospitalizations | 24 months |
| Number of major cardiovascular events and strokes (MACCE: death/myocardial infarction/revascularization /stroke) separately and combined | Number of cardiovascular<br>events and strokes (MACCE:<br>death/myocardial<br>infarction/revascularization<br>/stroke) | 24 months |
| Homeostatic Model Change<br>Assessment – Insulin<br>Resistance (HOMA-IR). | Homeostatic Model Assessment – Insulin Resistance (HOMA-IR) Change. | 12-24<br>months |
| Evaluation of change in the concentration of selected oxidative stress markers | Change in concentration of selected oxidative stress markers: catalase, superoxide dismutase (SOD), Oxygen Radical Absorbance Capacity (ORAC), total antioxidant capacity (TAC) | 12-24<br>months |





| Results | The study will evaluate the effect of treatment with flozin vs. semaglutide compared to treatment with metformin on the progression/regression of coronary atherosclerosis, change in plaque character, and control of cardiovascular risk factors in patients with non-obstructive coronary artery disease and pre-diabetic status |
|---|---|
| Interventions: | |
| Tested | Dapagliflozin (Forxiga), 10 mg film-coated tablets, oral |
| medicinal | |
| product #1 | |
| Tested drug | Semaglutide (Rybelsus), 3 mg tablets, 7 mg tablets, 14 mg tablets (target |
| product #2 | dose), oral |
| Other | Dietary, anti-smoking and appropriate physical activity counseling |
| interventions | |
| Comparator | Metformin (Formetic), 500 mg film-coated tablets or 1000 mg film-coated tablets, oral |
| Study schedule | Month and year of inclusion of the first participant: June 2024 |
| | Month and year of completion of the last participant's participation: |
| | June 2028 |
| | A pictorial diagram of the study is shown in Figure 1. A detailed schedule |
| | of appointments is provided in Section 8.6 (Table 1). |



Figure 1. Study diagram overview by appointments



# **Detailed schedule of appointments**

| Appointment | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time window (D-Day/W-Week/M- Month) | D0 | W2<br>(±3<br>D) | M1<br>(±3<br>D) | W6<br>(±3<br>D) | M2<br>(±3<br>D) | M6<br>(±3<br>D) | M9<br>(±3<br>D) | M12<br>(±9D<br>) | M15<br>(±9D<br>) | M18<br>(±9D<br>) | M21<br>(±9D<br>) | M24<br>(±9D<br>) |
| Clinical (K) /<br>Prescription (R) /<br>Telephone (T). | К | Т | К | т | К | К | R | К | R | К | R | К |
| Cardiology consultation | • | | • | | • | • | | • | | • | | • |
| Physical examination | • | | • | | • | • | | • | | • | | • |
| Presenting the patient with an offer to participate in the study. Discussing the risks and procedures involved in participating in the study. Providing the patient with an informed consent form for participation in the study | • | | | | | | | | | | | |
| Obtaining consent to participate in the study | • | | | | | | | | | | | |



| Performing an ECG | • | | | • | • | • | • |
|---|---|---|---|---|---|---|---|
| Collection of blood for determination of blood count, creatinine/GFR, lipid profile, glucose, Hba1c, insulin, lipoprotein A, ALT, AST, determination of TSH in selected patients (appointment V12); determination of hsCRP, HOMA-IR oxidative stress markers (appointment V1, V8, V12) | | • | • | • | • | • | • |
| General urinalysis | • | • | • | • | • | • | • |
| Taking measurements of weight, height, blood pressure, body composition, abdominal/hip circumference measurements | • | • | • | • | • | • | • |
| Assessment of comorbidities, diet (history) | • | • | • | • | • | • | • |
| Assessment of physical activity levels (e.g., using an app that measures physical activity levels on the patient's smartphone or other mobile device) | • | • | • | • | • | • | • |
| Advice on dietary | • | • | • | • | • | • | |



| | Π | | I | 1 | I | ı | Π | I | I | ı | 1 | I |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| goals and how to achieve them | | | | | | | | | | | | |
| Advice on optimizing physical activity levels | • | | • | | • | • | | • | | • | | |
| Advice on how to quit smoking | • | | | | | | | | | | | |
| Quality-of-life<br>assessment – EQ5D-<br>5L,Seattle Angina<br>Questionnaire <del>,</del> | • | | • | | • | • | | • | | • | | • |
| Randomization — allocation to the arm (experimental or control, 2:1) and, in the case of the experimental arm, to the appropriate drug group (flozin or semaglutide, 1:1), dispensing of the drug by support staff | • | | | | | | | | | | | |
| Transfer of CT imaging data records to the central imaging laboratory (Core Lab) for independent analysis | • | | | | | | | | | | | • |
| Evaluation of the occurrence of endpoints (according to the description of endpoints, Chapter 6) | | • | • | • | • | • | • | • | • | • | • | • |
| Collection of packages of drugs assigned during the previous appointment. Dispensing of new | | | • | | • | • | | • | | • | | • |



| drugs (except V12) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment of the regularity of the patient's drug intake | | • | • | • | • | • | • | • | • | • | • | • |
| Evaluation of the tolerability of the assigned drugs, taking into account potential side effects | | • | • | • | • | • | • | • | • | • | • | • |
| Reminder to follow dietary recommendations and maintain adequate levels of physical activity | | • | | • | | | • | | • | | • | |
| Pregnancy test | • | | | | | | | | | | | • |
| Coronary CT study | | | | | | | | | | | | • |
| Providing recommendations for treatment after participation in the study | | | | | | | | | | | | • |

Table 1. Detailed scope of activities and procedures performed during appointments